CLINICAL TRIAL: NCT04865757
Title: Space Flap for Cerebral Protection Following Decompressive Hemicraniectomy for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080/12
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Infarction
Keywords: Decompressive hemi-craniectomy; bone flap
MeSH Terms: conditions — Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Space Flap (Experimental): A space flap is formed out of Palacos®, adjusted to the skull surface with temporal augmentation
  Interventions: Device: Space Flap

INTERVENTIONS:
Device: Space Flap — A space flap is formed out of Palacos®, adjusted to the skull surface with temporal augmentation

SUMMARY:
In this study the investigators want to investigate to what extent the application of an artificial bone flape (space flap) influences the success of a decompressive craniectomy.

In all participants, a space flap is placed immediately after removal of the skull cap. In a second operation, after 1-3 months, an operation is performed, in which the stored own skull bone is re-inserted. The artificial bone cover is removed at this point.

DETAILED DESCRIPTION:
The destruction of local brain parenchyma after cerebral infarction leads to local swelling within a few days. In the beginning the ischemic brain expand at the expense of the CSF and venous spaces. However, once these spaces are partially displaced further swelling invariably leads to increase of the intracranial pressure due to the limited space available inside the cranial vault. In cases of large infarctions this increase in intracranial pressure (ICP) may entail life threatening secondary injuries to the brain. The surgical removal of a large part of the skull (decompressive hemi-craniectomy) allows the ischemic brain to expand, therefore avoiding an increase of ICP and it's deleterious effects. After removal of a part of the skull the skin is closed again, and the skull flap is kept in sterile environment. Several months after decompression craniectomy patients undergo implantation of either their preserved bone flap or of a bone flap substitute (so-called patient specific implant, or PSI, mostly made out of Palacos®).

Decompressive hemi-craniectomy comes at a cost for the patient, despite its undisputed role as a life saving surgery after large cerebral infarction. During the first days after surgery the brain may use the space freed up by bone removal. In some cases the brain may prolapse even further out of the cranial vault, leading to brain herniation. Brain herniation are common and may lead to further damage due to axonal shearing injuries in the brain, and to hemorrhages and infarction at the craniotomy edges. The lack of the protective skull prior to re-implantation of the bone flap puts the brain at risk of injuries due to falls during rehabilitation and exposes the brain indirectly to atmospheric pressure. Various neurological deficits subsumed as the syndrome of the trephined have been described in these patients. The symptoms of the syndrome of the trephined have in common that they appear a few weeks after decompression and significantly improve after re-implantation of the patient's own bone. The symptoms range from orthostatic headache and dizziness to motor paresis, aphasia, cognitive decline and brainstem compression symptoms. The pathophysiology behind the syndrome of the trephined can be understood as an "open box" phenomenon. After removal of the bone the brain is separated from the atmospheric pressure only by the skin. The skin, however, does not hold against atmospheric pressure and sinks into the skull cavity (sinking skin flap) once the brain swelling diminishes. Physiologic dynamics of the cerebrospinal fluid are deranged, leading to hydrocephalus, subdural hygromas and parenchymal effusions. This assumption is enforced by pathophysiological observations of decreased cerebral blood flow in both hemispheres following decompression, and normalization thereof following re-implantation of the bone flap.

This pilot study aims at assessing feasibility of a change in surgical protocol. The rate of ICP control will be used to determine the sample size of a planned monocenter study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Decompressive hemi-craniectomy planed for*:

  * Impairment of consciousness or progressive reduction of consciousness and
  * Mass effect on brain imaging (oedema exceeding 50% of the MCA territory and midline shift), and
  * Exclusion of other causes of impaired consciousness (e.g. hypoperfusion, hypotension, cerebral reinfarction, epileptic seizures
* Informed consent from relatives

Exclusion Criteria:

* Bilateral, nonreactive, not drug-induced pupillary dilation, associated with coma*
* Simultaneous presence of all four of the following unfavorable prognostic factors: *

  * Age 50 years
  * Involvement of additional vascular territories
  * Unilateral pupillary dilation
  * GCS<8
* Severe comorbidity (severe heart failure or myocardial infarction, incurable neoplasia, etc. *
* Refusal by the patient of this treatment, as known from current interaction with the patient, from existing written documents or related by the patient's proxies. *
* Known pulmonary or cranial infection
* Any coagulopathy
* Rapid neurological decline prohibiting the extra time needed for space flab production (10min)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
ICP Control | 1 day after surgery
  ICP Control (number of hours with mean ICP equal to or > 20mmHg)

SECONDARY OUTCOMES:
Intracranial infections | 1 day after surgery
  Intracranial infections (proven by microbiology)
Postoperative hematomas | 1 day after surgery
  Postoperative hematomas localized at the edge of the craniotomy
Postoperative infarctions | 1 day after surgery
  Postoperative infarctions localized at the edge of the craniotomy
Brain herniation | 1 day after surgery
  Brain herniation (>1.5cm out of cranial vault)
Syndrom of the trephined | 1 day after surgery
  Syndrom of the trephined assessed by MRI/CT Scan
Hydrocephalus malresorptivus | 1 month after surgery
  Hydrocephalus malresorptivus assessed by MRI/CT Scan
Adhesions between the brain and the skin | 1 month after surgery
  Adhesions between the brain and the skin
Adhesions between the palacos and the temporal muscle | 1 month after surgery
  Adhesions between the palacos and the temporal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Schucht Philippe, MD, Principal Investigator — Dep. of Neurosurgery, Bern University Hospital
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Langfitt TW. Increased intracranial pressure. Clin Neurosurg. 1969;16:436-71. doi: 10.1093/neurosurgery/16.cn_suppl_1.436. No abstract available. PMID 4981573
- [Background] Steiger HJ. Outcome of acute supratentorial cerebral infarction in patients under 60. Development of a prognostic grading system. Acta Neurochir (Wien). 1991;111(3-4):73-9. doi: 10.1007/BF01400491. PMID 1950691
- [Background] Wirtz CR, Steiner T, Aschoff A, Schwab S, Schnippering H, Steiner HH, Hacke W, Kunze S. Hemicraniectomy with dural augmentation in medically uncontrollable hemispheric infarction. Neurosurg Focus. 1997 May 15;2(5):E3; discussion 1 p following E3. doi: 10.3171/foc.1997.2.5.7. PMID 15096004
- [Background] Doerfler A, Engelhorn T, Forsting M. Decompressive craniectomy for early therapy and secondary prevention of cerebral infarction. Stroke. 2001 Mar;32(3):813-5. doi: 10.1161/01.str.32.3.813. No abstract available. PMID 11239209
- [Background] Juttler E, Schwab S, Schmiedek P, Unterberg A, Hennerici M, Woitzik J, Witte S, Jenetzky E, Hacke W; DESTINY Study Group. Decompressive Surgery for the Treatment of Malignant Infarction of the Middle Cerebral Artery (DESTINY): a randomized, controlled trial. Stroke. 2007 Sep;38(9):2518-25. doi: 10.1161/STROKEAHA.107.485649. Epub 2007 Aug 9. PMID 17690310
- [Background] Hofmeijer J, Kappelle LJ, Algra A, Amelink GJ, van Gijn J, van der Worp HB; HAMLET investigators. Surgical decompression for space-occupying cerebral infarction (the Hemicraniectomy After Middle Cerebral Artery infarction with Life-threatening Edema Trial [HAMLET]): a multicentre, open, randomised trial. Lancet Neurol. 2009 Apr;8(4):326-33. doi: 10.1016/S1474-4422(09)70047-X. Epub 2009 Mar 5. PMID 19269254
- [Background] Vahedi K, Vicaut E, Mateo J, Kurtz A, Orabi M, Guichard JP, Boutron C, Couvreur G, Rouanet F, Touze E, Guillon B, Carpentier A, Yelnik A, George B, Payen D, Bousser MG; DECIMAL Investigators. Sequential-design, multicenter, randomized, controlled trial of early decompressive craniectomy in malignant middle cerebral artery infarction (DECIMAL Trial). Stroke. 2007 Sep;38(9):2506-17. doi: 10.1161/STROKEAHA.107.485235. Epub 2007 Aug 9. PMID 17690311
- [Background] Sanus GZ, Tanriverdi T, Ulu MO, Kafadar AM, Tanriover N, Ozlen F. Use of Cortoss as an alternative material in calvarial defects: the first clinical results in cranioplasty. J Craniofac Surg. 2008 Jan;19(1):88-95. doi: 10.1097/scs.0b013e31815c93fe. PMID 18216670
- [Background] Wagner S, Schnippering H, Aschoff A, Koziol JA, Schwab S, Steiner T. Suboptimum hemicraniectomy as a cause of additional cerebral lesions in patients with malignant infarction of the middle cerebral artery. J Neurosurg. 2001 May;94(5):693-6. doi: 10.3171/jns.2001.94.5.0693. PMID 11354398
- [Background] Honeybul S, Ho KM. Long-term complications of decompressive craniectomy for head injury. J Neurotrauma. 2011 Jun;28(6):929-35. doi: 10.1089/neu.2010.1612. Epub 2011 Jun 1. PMID 21091342
- [Background] Aarabi B, Hesdorffer DC, Ahn ES, Aresco C, Scalea TM, Eisenberg HM. Outcome following decompressive craniectomy for malignant swelling due to severe head injury. J Neurosurg. 2006 Apr;104(4):469-79. doi: 10.3171/jns.2006.104.4.469. PMID 16619648
- [Background] Sakamoto S, Eguchi K, Kiura Y, Arita K, Kurisu K. CT perfusion imaging in the syndrome of the sinking skin flap before and after cranioplasty. Clin Neurol Neurosurg. 2006 Sep;108(6):583-5. doi: 10.1016/j.clineuro.2005.03.012. PMID 15921849
- [Background] Dujovny M, Fernandez P, Alperin N, Betz W, Misra M, Mafee M. Post-cranioplasty cerebrospinal fluid hydrodynamic changes: magnetic resonance imaging quantitative analysis. Neurol Res. 1997 Jun;19(3):311-6. doi: 10.1080/01616412.1997.11740818. PMID 9192385
- [Background] Stiver SI, Wintermark M, Manley GT. Reversible monoparesis following decompressive hemicraniectomy for traumatic brain injury. J Neurosurg. 2008 Aug;109(2):245-54. doi: 10.3171/JNS/2008/109/8/0245. PMID 18671636
- [Background] Mokri B. Orthostatic headaches in the syndrome of the trephined: resolution following cranioplasty. Headache. 2010 Jul;50(7):1206-11. doi: 10.1111/j.1526-4610.2010.01715.x. Epub 2010 Jun 18. PMID 20561067
- [Background] Joseph V, Reilly P. Syndrome of the trephined. J Neurosurg. 2009 Oct;111(4):650-2. doi: 10.3171/2009.3.JNS0984. PMID 19361266
- [Background] Bijlenga P, Zumofen D, Yilmaz H, Creisson E, de Tribolet N. Orthostatic mesodiencephalic dysfunction after decompressive craniectomy. J Neurol Neurosurg Psychiatry. 2007 Apr;78(4):430-3. doi: 10.1136/jnnp.2006.099242. Epub 2006 Nov 21. PMID 17119005
- [Background] Akins PT, Guppy KH. Sinking skin flaps, paradoxical herniation, and external brain tamponade: a review of decompressive craniectomy management. Neurocrit Care. 2008;9(2):269-76. doi: 10.1007/s12028-007-9033-z. PMID 18064408
- [Background] Fodstad H, Love JA, Ekstedt J, Friden H, Liliequist B. Effect of cranioplasty on cerebrospinal fluid hydrodynamics in patients with the syndrome of the trephined. Acta Neurochir (Wien). 1984;70(1-2):21-30. doi: 10.1007/BF01406039. PMID 6741628
- [Background] Yang XF, Wen L, Shen F, Li G, Lou R, Liu WG, Zhan RY. Surgical complications secondary to decompressive craniectomy in patients with a head injury: a series of 108 consecutive cases. Acta Neurochir (Wien). 2008 Dec;150(12):1241-7; discussion 1248. doi: 10.1007/s00701-008-0145-9. Epub 2008 Nov 13. PMID 19005615
- [Background] Won YD, Yoo DS, Kim KT, Kang SG, Lee SB, Kim DS, Hahn ST, Huh PW, Cho KS, Park CK. Cranioplasty effect on the cerebral hemodynamics and cardiac function. Acta Neurochir Suppl. 2008;102:15-20. doi: 10.1007/978-3-211-85578-2_3. PMID 19388280
- [Background] Michel P, Arnold M, Hungerbuhler HJ, Muller F, Staedler C, Baumgartner RW, Georgiadis D, Lyrer P, Mattle HP, Sztajzel R, Weder B, Tettenborn B, Nedeltchev K, Engelter S, Weber SA, Basciani R, Fandino J, Fluri F, Stocker R, Keller E, Wasner M, Hanggi M, Gasche Y, Paganoni R, Regli L; Swiss Working Group of Cerebrovascular Diseases with the Swiss Society of Neurosurgery and the Swiss Society of Intensive Care Medicine. Decompressive craniectomy for space occupying hemispheric and cerebellar ischemic strokes: Swiss recommendations. Int J Stroke. 2009 Jun;4(3):218-23. doi: 10.1111/j.1747-4949.2009.00283.x. No abstract available. PMID 19659825